CLINICAL TRIAL: NCT05055076
Title: Retrospective Study to Investigate Rotational Stability and Clinical Outcomes After Implantation of a Monofocal Toric Intraocular Lens (IOL)
Brief Title: PMCF Retrospective Study Outcomes of a Monofocal Toric Intraocular Lens
Status: Completed | Type: Observational
Sponsor: Beaver-Visitec International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PHY2120
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Cataract; Lens Opacities; Astigmatism
Keywords: Intraocular Lens; Monofocal; Toric Lens
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PODEYE TORIC: Adult patients who have undergone cataract surgery with mono- or bilateral implantation of POD EYE TORIC IOL (POD T 49P) and who meet all the inclusion and exclusion criteria will be invited to participate in the study.
  Interventions: Device: PODEYE TORIC

INTERVENTIONS:
Device: PODEYE TORIC — Patients will be contacted consecutively and will be enrolled after the patient informed leaflet has been given to them and after obtaining their consent to the scientific use of their data collected retrospectively (preoperative, surgery, postoperative routine visits). Patients will only be enrolled after the routine 4-6 months visit has been performed.

SUMMARY:
This is a monocentric retrospective, open-label clinical study in patients after unilateral or bilateral implantation of hydrophobic acrylic monofocal toric intraocular lens PODEYE TORIC and executed only with standard of care examinations.

The investigational device is CE approved. The investigational device and all study products, including the devices used for the study examinations, have been used within the intended use specifications from the manufacturer. In addition, there were no invasive or other burdening examinations.

The investigator is an accredited and experienced cataract surgeon and researcher.

The primary endpoint is to determine rotational stability in a minimum of 120 eyes of patients with PODEYE TORIC IOL implantation after cataract surgery. Patients will be enrolled for the documentation and evaluation of retrospective data up to 6 months postoperatively.

DETAILED DESCRIPTION:
Age-related changes of the proteins in the crystalline lens lead to cataract formation. Cataracts are a common condition in adults over 40 years of age, and surgical replacement of the cataractous lens with an intraocular lens (IOL) remains an effective way to restore vision to cataract patients.

On patients with a low amount of pre-existing corneal astigmatism (defect in the sphericity of the cornea with a focal point depending on the meridian), the implantation of a spherical monofocal IOL is the state- of- the-art when targeting a good correction of distance visual function. However, in case of pre-existing corneal astigmatism, the implantation of spherical IOLs might not be the best solution, as such lenses only correct for spherical errors and leave the astigmatism uncorrected.

Toric IOLs are obtained by adding a cylinder power to the basis optic of a given spherical power, thus correcting for both spherical and cylindrical refractive errors. Toric IOLs provide the opportunity to reduce or eliminate astigmatism, thus offering patients with pre-existing astigmatism the possibility of restoring their distance vision with reduced or no need for the use of spectacles or contact lenses with a cylindrical correction. Not correcting the astigmatism component at the time of cataract surgery is an important cause for not obtaining planned emmetropia following IOL implantation. A previous study found that more than 22% of patients undergoing cataract surgery have substantial corneal astigmatism superior than 1.25 D and would benefit from toric IOL implantation 1).

This study will add to the knowledge on toric IOLs and help improve the care of patients and the outcomes of cataract surgery after toric IOL implantation.

The study is a monocentric, retrospective study to investigate rotational stability and visual performance after mono- or bilateral implantation of PODEYE TORIC intraocular lens following cataract surgery, executed only with standard of care examinations. The study outcomes will be used to confirm the safety performance for a stable IOL positioning of the investigation al device.

Preoperative, surgical and postoperative data (up to 6 months after surgery) will be collected retrospectively by reviewing the patient charts.

The investigational device PODEYE TORIC IOL is CE approved and commercially available in the country where this clinical investigation is being carried out. The investigational device and all study products, including the devices used for the study examinations, have been used within the intended use specifications from the manufacturer. In addition, no invasive or other burdening examinations will occur for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged 35 years or older on the day of treatment that were mono- or bilaterally implanted with PODEYE TORIC intraocular lens
* Capable of understanding the patient informed leaflet;
* Complete data available at the screening visit, surgical visit and at least one postoperative visit.

Exclusion Criteria:

* Age of patient <35 years at the day of surgery;
* Subjects who underwent previous intraocular or corneal surgery other than IO L implantation;
* Subjects in whom in-the-bag implantation was not possible;
* Subjects in whom surgical complications occurred (e.g. posterior rupture);

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have undergone cataract surgery with mono- or bilateral implantation of POD EYE TORIC IOL (POD T 49P) and who meet all the inclusion and exclusion criteria will be invited to participate in the study.
  Patients will be contacted consecutively and will be enrolled after the patient informed leaflet has been given to them and after obtaining their consent to the scientific use of their data collected retrospectively (preoperative, surgery, postoperative routine visits). Patients will only be enrolled after the routine 4-6 months visit has been performed.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Rotational Stability | 6 months
  Rotational stability is an important parameter on toric IOLs, as postoperative IO L rotation can lead to inappropriate correction of corneal astig matism and decrease in uncorrected distance visual acuity.
  The primary study endpoint is the absolute value of rotation between the day of surgery and the postoperative visit 6 months after surgery. The absolute value of rotation should be less than 10° in 90% of the eyes implanted with POD EYE TORIC lens according to safety declarations of EN ISO 11979-7:2018.

SECONDARY OUTCOMES:
Stability of Manifest Refraction (Spherical Equivalent) | 6 months
  Manifest refraction will be assessed using the spherical equivalent: Manifest refraction Spherical
  Equivalent (MRSE). Negative cylinder notation will be used. MRSE is calculated by the following formula:
  MRSE = sphere + 1/2 cylinder. Descriptive analysis of sphere, cylinder and MRS E will be reported. Stability of the MRSE will be assessed by summarizing the change in MRSE between adjacent visits ( mean, standard deviation, minimum and maximum, and 95% confidence interval).

OTHER OUTCOMES:
Corrected and Uncorrected Distance Visual Acuity | 6 months
  Corrected and Uncorrected Distance Visual Acuity data will be measured and summarized (mean, standard deviation, minimum and maximum) at each visit, as far as available, and the change between visits with a 95% confidence interval will be provided.
Refractive astigmatism predictability | 6 months
  The refractive astig matism predictability achieved with the PhyslO L toric calculator will be assessed and compared to other toric calculators. The prediction error will be calculated as the difference between the measured postoperative manifest refraction and the predicted residual astigmatism.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Beau Soleil, Montpellier, France

IPD SHARING:
Plan to Share IPD: No